CLINICAL TRIAL: NCT03111251
Title: Multi-component Interventions for Patients and Providers to Increase HPV Vaccination in a Network of Pediatric Clinics in Houston, TX
Brief Title: Multi-component Interventions to Increase HPV Vaccination in a Network of Pediatric Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other); Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Sally Vernon, ◦Blair Justice, PhD Professorship in Mind-Body Medicine and Public Health and Director, Division of Health Promotion and Behavioral Sciences, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-15-0202
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Human Papillomavirus (HPV)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Provider-only intervention (Experimental): New provider- and system-level evidence-based strategies for increasing HPV vaccination rates are being implemented throughout the entire clinic network. This includes provider assessment and feedback, provider reminders, provider education, and patient reminders.
  Interventions: Behavioral: Provider assessment and feedback; Behavioral: Provider reminders; Behavioral: Provider education; Behavioral: Patient reminders
- Provider plus parent intervention (Experimental): Clinics randomized to the provider plus parent intervention will receive both the provider intervention and the parent education intervention.
  Interventions: Behavioral: Provider assessment and feedback; Behavioral: Provider reminders; Behavioral: Provider education; Behavioral: Patient reminders; Behavioral: Parent education

INTERVENTIONS:
Behavioral: Provider assessment and feedback — Tailored immunization reports highlighting adolescent vaccination rates at the individual, clinic and network levels are distributed by clinic champions every quarter. Reports track vaccination rates over time and allow physicians to compare their rates to the national goal.
Behavioral: Provider reminders — An EHR-based reminder system informs providers when patients are due or overdue for HPV vaccination.
Behavioral: Provider education — Provider education is being delivered through a comprehensive online continuing education activity that is tailored specifically to physicians, nurses, and clinical staff at TCP practices. It focuses on HPV vaccination best practices and communicating with parents about the HPV vaccine.
Behavioral: Patient reminders — Patient reminders are delivered through MyChart, the clinics' online personal health record system, to inform patients (parents) that they are due or overdue for HPV vaccination.
Behavioral: Parent education — The parent education intervention (currently in development) will employ innovative strategies to identify and overcome barriers to HPV vaccination.
  Arms: Provider plus parent intervention

SUMMARY:
The purpose of the study is to determine the comparative effectiveness of a provider-only intervention and a parent plus provider intervention to increase initiation of HPV vaccination among male and female patients ages 11-17 in a large pediatric clinic network in the greater Houston area. The hypothesis is that HPV vaccine initiation will be higher in clinics randomized to the parent plus provider intervention compared with clinics randomized to the provider-only intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patient at a Texas Children's Pediatrics clinic
* Patient had not initiated the HPV vaccination series at baseline

Exclusion Criteria:

- Patient had completed the HPV vaccination series at baseline

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2015-03-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Change in percent of HPV vaccination initiation | baseline, 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Sally W Vernon, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States